CLINICAL TRIAL: NCT07089199
Title: Tislelizumab Combined With Anlotinib and Nab-paclitaxel in III Resectable Non-small Cell Lung Cancer : A Prospective, Single-Arm, Phase II Study
Brief Title: Tislelizumab Combined With Anlotinib and Nab-paclitaxel in III Resectable Non-small Cell Lung Cancer(TitAN) : A Prospective, Single-Arm, Phase II Study
Acronym: TitAN
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KYLL-202406-009-1
Record Dates: First submitted 2025-07-20; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: NSCLC; Tislelizumab; Anlotinib; Nab-paclitaxel
MeSH Terms: interventions — Neoadjuvant Therapy; Surgical Procedures, Operative; Chemotherapy, Adjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- treatment arm (Experimental): Participants received 3-4 cycles of Tislelizumab combined with anlotinib and nab-paclitaxel treatment, once every 3 weeks, for a maximum of 4 cycles.
  Patients who meet the surgical conditions will undergo surgery within 4 to 6 weeks after neoadjuvant therapy.
  After the operation, the patient entered the stage of single-agent adjuvant therapy with tislelizumab. The adjuvant therapy with tislelizumab lasted for one year (including preoperative treatment medication, a total of 17 cycles)
  Interventions: Drug: neoadjuvant therapy; Procedure: Surgery; Drug: Adjuvant therapy

INTERVENTIONS:
Drug: neoadjuvant therapy — tislelizumab （200mg，iv, q3w） + Anlotinib （10mg, orally, D1-14, q3w）+nab-paclitaxel（260mg/m2，q3w）3-4cycle
Procedure: Surgery — Surgery should be performed 4 to 6 weeks after the last neoadjuvant therapy (at least 4 weeks after the end of anlotinib treatment).
Drug: Adjuvant therapy — Tislelizumab: 200mg, iv, Q3W, 1year at most(including preoperative treatment medication, a total of 17 cycles).

SUMMARY:
This study is a single-arm prospective clinical trial. The primary objective of the study is to explore the efficacy and safety of preoperative neoadjuvant therapy with Tislelizumab combined with Anlotinib and Nab-Paclitaxel in resectable stage III non-small cell lung cancer.Finally, it provides new evidence-based medical evidence for the perioperative treatment of non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years old, gender is not limited;
2. Histologically confirmed Stage III non-small cell lung cancer (AJCC Stage 8th edition)
3. The tumor is resectable after assessment by the attending surgeon
4. EGFR/ALK mutation negative or unknown (unknown only for squamous non-small cell lung cancer)
5. Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
6. No previous treatment received
7. At least 1 measurable lesion as defined by RECIST v1.1
8. Be able to provide the Informed Consent Form (ICF), and be able to understand and agree to abide by the research requirements and assessment schedule
9. Good organ function; • Patients have not received blood transfusion or growth factor support therapy ≤ 14 days prior to sample collection during the screening period and: Absolute neutral cell count (ANC) ≥1.5 x 109/L Platelet ≥100 x 109/L Hemoglobin ≥90 g/L • Calculated creatinine clearance (CrCl) (Cockcroft-Gault formula) creatinine clearance ≥ 45 mL/min Serum total bilirubin ≤1.5 × upper limit of normal (ULN) (patients with Gilbert's syndrome must have total bilirubin < 3 × ULN) AST and ALT≤ 2.5 x ULN Patients who did not receive anticoagulant therapy: International standardized ratio or activated partial thromboplastin time ≤ 1.5 × ULN
10. Women of childbearing age must take a serum pregnancy test within 3 days before the first medication, and the result is negative. Female subjects of reproductive age and male subjects whose partners are women of reproductive age must agree to use highly effective methods of contraception during the study period and for 120 days after the last dose of the study drug

Exclusion Criteria:

1. A history of received treatment for current lung cancer, including radiotherapy and all systemic antitumor agents, including chemotherapy, immunotherapy, targeted therapy or antiangiogenic therapy.
2. Patients with known EGFR gene mutation, ALK rearrangement, ROS-1 fusion, RET fusion, HER-2 mutation, MET mutation, but if patients with squamous non-small cell lung cancer, the EGFR mutation status and ALK mutation status are unknown, it is not required to conduct tests during screening
3. There are multiple factors influencing patients taking oral medication (such as inability to swallow, chronic diarrhea, intestinal obstruction)
4. Allergy to any study drug (Tislelizumab, Anlotinib, albumin-bound Paclitaxel) or excipients.
5. Imaging shows that the tumor has invaded important blood vessels or the investigator judges that the tumor invasion of important blood vessels during treatment is likely to cause fatal bleeding.
6. Clinically significant hemoptysis (more than 50 ml per day) within 3 months before the study, or clinically significant bleeding symptoms or obvious bleeding tendency (such as gastrointestinal bleeding, gastric ulcer bleeding, gastrointestinal bleeding, hemorrhagic gastric ulcer, fecal occult blood ++ and above baseline, or suffering from vasculitis, etc.).
7. Vaccination with attenuated live vaccines within 4 weeks before the first dose or planned vaccination during the study period.
8. Patients who are expected to be unable to tolerate surgery, such as those with cardiopulmonary insufficiency.
9. Occurrence of or concurrent other malignancies within the past 5 years, except for cured cervical carcinoma in situ, non-melanoma skin cancer, and superficial bladder tumors [Ta (non-invasive tumor), Tis (carcinoma in situ), and T1 (tumor invading the basement membrane)].
10. Patients with active viral hepatitis requiring treatment as determined by the investigator.
11. Active autoimmune diseases requiring systemic treatment, or long-term use of high doses of steroids or other immunomodulators, which the investigator assesses as affecting the study treatment.
12. Unhealed surgical incisions before the start of study treatment (small biopsy incisions can be included).
13. Active hepatitis B/C infection and human immunodeficiency virus (HIV) infection.
14. Arterial or venous thrombotic events within 6 months (such as cerebrovascular accident, deep vein thrombosis, pulmonary embolism, etc.) or severe cardiovascular diseases: myocardial ischemia or myocardial infarction above grade II, uncontrolled arrhythmias; heart failure above grade III-IV according to NYHA standards, or left ventricular ejection fraction (LVEF) < 50% as indicated by echocardiography.
15. Interstitial lung disease, uncontrolled systemic medical history, including diabetes, hypertension, acute lung disease, etc.
16. Active bleeding or coagulation dysfunction (INR > 2.0, PT > 16s), bleeding tendency or receiving thrombolytic, anticoagulant, antiplatelet therapy; any major surgery requiring general anesthesia within ≤ 28 days before the first dose.
17. Underlying medical conditions or alcohol/drug abuse that are unfavorable for the administration of study drugs, may affect the interpretation of results, or pose a high risk of treatment complications.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-07-25 (Estimated); Primary Completion 2026-07-10 (Estimated); Study Completion 2028-07-10 (Estimated)

PRIMARY OUTCOMES:
pathological complete response (pCR) | Up to approximately 8 weeks following completion of neoadjuvant treatment
  pCR rate is defined as the percentage of participants having an absence of residual invasive cancer in resected lung specimens and lymph nodes following completion of neoadjuvant therapy.

SECONDARY OUTCOMES:
Major Pathological Response (mPR) Rate | Up to approximately 8 weeks following completion of neoadjuvant treatment
  mPR rate is defined as the percentage of participants having ≤10% viable tumor cells in the resected primary tumor and all resected lymph nodes following completion of neoadjuvant therapy.
R0 resection rate | usually 1 week after surgery
  R0 Resection Rate: The pathological results will showed that the incision margin was negative and no residual cancer cells were found under the microscope.
Event-Free Survival(EFS) | Up to 2years
  The time from the start of randomization (or the start of treatment in a one-arm trial) to the first occurrence of any of the following events: disease progression without surgical treatment, local or distant recurrence, death from any cause, etc.
overall survival(OS) | 3 years
  Time from randomization to death (from any cause)
Safety and Tolerability | Up to 3 years
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0

IPD SHARING:
Plan to Share IPD: Undecided